CLINICAL TRIAL: NCT01047657
Title: Effects of Weight Loss in Obese Difficult-to-treat Asthmatics: a Pilot Study
Brief Title: Effects of Weight Loss in Obese Difficult-to-treat Asthmatics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Alberto Cukier, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBSTRUÇÃOHC-01
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2009-12

CONDITIONS: Asthma; Obesity; Weight Loss
Keywords: Asthma; Obesity; weight loss
MeSH Terms: conditions — Asthma; Obesity; Weight Loss | interventions — Caloric Restriction; Orlistat; sibutramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- weight loss (Experimental)
  Interventions: Behavioral: Low caloric diet plus orlistat and sibutramine
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Low caloric diet plus orlistat and sibutramine — All subjetcs
  Arms: weight loss

SUMMARY:
Sixty percent of patients with difficult to control asthma seen in our outpatient clinic are obese. The impact of weight reduction in this subpopulation of asthmatics has not been studied. Our aim is to evaluate the impact of weight reduction on asthma control of these patients.

DETAILED DESCRIPTION:
Study design: interventional, open label, randomized

Patients selection

Thirty-three difficult to control obese asthmatic patients, aged between 18 to 65 years old will be recruited from the outpatient clinics of the Pulmonary Division of the University of Sao Paulo Hospital.

Difficult to control asthma will be defined as patients who do not achieve asthma control (according to GINA) despite best treatment regimen and checked adherence after at least three months of treatment.

Intervention: Patients will be divided in two groups: asthma treatment plus weight loss program or asthma treatment alone for 6 months without drug dose changing.

Procedures (baseline and after 6 months) - quality of life questionnaire, asthma control questionnaire, lung function tests, serum and sputum inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Difficult-to-treat asthma
* Body mass index > 30kg/m2

Exclusion Criteria:

* Subjets older than 65 years
* Current smoking
* Past smoking history (> 10 pack-year)
* Pregnancy
* Contraindication for Orlistat or Sibutramine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Asthma control questionnaire (ACQ) | Baseline and six months

SECONDARY OUTCOMES:
Inflammatory parameters | Baseline and after 6 months
Pulmonary mechanics | Baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sérvulo A. Dias-Júnior, MD, Principal Investigator — Heart Institute, University of São Paulo; Alberto Cukier, PhD, Study Director — Heart Institute, University of São Paulo
Locations (1):
- University of São Paulo - Heart Institute and Hospital das Clínicas, São Paulo, São Paulo, Brazil